CLINICAL TRIAL: NCT05769881
Title: The Effects of Subcostal Transversus Abdominis Plane Block and Local Anesthetic Infiltration on Post-operative Stress Hormone and Pain Relief After Laparoscopic Cholecystectomy
Brief Title: Effects of Subcostal TAP Block and Local Anesthetic Infiltration After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ilay Cetiner, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1221
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain; Subcostal Transversus Abdominis Plane Block; Gall Bladder Disease
Keywords: Cholecystectomy, Laparoscopic; Subcostal Transversus Abdominis Plane Block; Analgesia; Cortisol; Prolactin
MeSH Terms: conditions — Pain, Postoperative; Gallbladder Diseases; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided subcostal transversus abdominis plane block (Active Comparator): After the induction of anesthesia, before the beginning of the operation, the subcostal transversus abdominis region is going to be detected under ultrasound guidance and 25-30 ml of 0.25% bupivacaine will be administered
  Interventions: Procedure: Ultrasound guided subcostal transversus abdominis plane block
- Wound site local anesthetic infiltration (Active Comparator): After induction of anesthesia, before the beginning of the operation, a total of 20 ml of 0.25% bupivacaine is going to be infiltrated in equal doses to the four regions that will have trocar access.
  Interventions: Procedure: Wound site local anesthetic infiltration

INTERVENTIONS:
Procedure: Ultrasound guided subcostal transversus abdominis plane block — After the induction of anesthesia, before the beginning of the operation, the subcostal transversus abdominis region is going to be detected under ultrasound guidance and 25-30 ml of 0.25% bupivacaine will be administered
  Arms: Ultrasound guided subcostal transversus abdominis plane block
Procedure: Wound site local anesthetic infiltration — After induction of anesthesia, before the beginning of the operation, a total of 20 ml of 0.25% bupivacaine is going to be infiltrated in equal doses to the four regions that will have trocar access
  Arms: Wound site local anesthetic infiltration

SUMMARY:
Laparoscopic cholecystectomy surgery is an intra-abdominal surgery that is frequently used in the treatment of gallbladder-related pathologies. Compared to open surgery, the cost, the risk of bleeding, the risk of surgical site infection are lower, the need for hospitalization is shorter, and the recovery is rapid. Adequate pain relief is very important after laparoscopic cholecystectomy. Inadequate analgesia in post-operative period has been associated with pain-related cognitive dysfunction, atelectasis, thromboembolic events, increased surgery-related stress response, prolonged hospital stay, and chronic pain in patients. Acetaminophen, non-steroidal anti-inflammatory drugs, opioid analgesics, intraperitoneal washing, local anesthesia infiltration and various regional anesthesia techniques can be used for appropriate analgesia. Studies have shown that subcostal transversus abdominis block has good analgesic efficacy in laparoscopic cholecystectomy surgeries. In the perioperative and postoperative period, afferent nerve signals in the surgical incision area stimulate the hypothalamus, causing the release of CRH, arginine vasopressin, and cortisol depending on the size of the surgical procedure. Providing patients with appropriate postoperative analgesia reduces the release of the stress hormones cortisol and prolactin.

In this study, the investigators are aiming to compare the post-operative analgesic affects and stress hormone responses of subcostal transversus abdominis plane block and local anesthetic infiltration in patients undergoing laparoscopic surgery. The study is planned to be prospective, randomized and single-blind.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy surgery is an intra-abdominal surgery that is frequently used in the treatment of gallbladder-related pathologies. With the widespread use of laparoscopic procedures, open surgery has been replaced by laparoscopic cholecystectomy. Compared to open surgery, the cost, the risk of bleeding, the risk of surgical site infection are lower, the need for hospitalization is shorter, and the recovery is rapid.

Post-abdominal pain is carried by T6-L1 thoracolumbar nerves. Pain after laparoscopic cholecystectomy has both visceral and parietal components, and patients are generally more bothered by visceral pain after surgery. Visceral pain arises from intraperitoneal inflammation and increases with coughing, respiratory effort, and mobilization in the post-operative period, and inadequate analgesia in this period has been associated with pain-related cognitive dysfunction, atelectasis, thromboembolic events, increased surgery-related stress response, prolonged hospital stay, and chronic pain in patients. Acetaminophen, non-steroidal anti-inflammatory drugs, opioid analgesics, intraperitoneal washing, local anesthesia infiltration and various regional anesthesia techniques can be used for appropriate analgesia. Studies have shown that subcostal transversus abdominis block has good analgesic efficacy in laparoscopic cholecystectomy surgeries.

In the perioperative and postoperative period, afferent nerve signals in the surgical incision area stimulate the hypothalamus, causing the release of CRH, arginine vasopressin, and cortisol depending on the size of the surgical procedure. Providing appropriate postoperative analgesia in patients decreased the release of stress hormones cortisol and prolactin.

In this study, the investigators are aiming to compare the effects of subcostal transversus abdominis block and local anesthetic infiltration on postoperative analgesia and stress hormone response in patients who underwent laparoscopic cholecystectomy surgery. The study is planned to be prospective, randomized and single-blind.

ELIGIBILITY:
Inclusion Criteria:

* who will undergo laparoscopic cholecystectomy
* ASA I-II
* 18-65 age group

Exclusion Criteria:

* Pregnant
* Emergency surgery
* ASA III-IV
* History of local anesthetic allergy
* Coagulative disorder
* Corticosteroid use
* Severe psychiatric disease
* History of chronic pain
* Uncooperative patients
* Neurological deficit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
VAS score | 24 hours
  Patients are going to be evaluated for 24 hours postoperatively with recording of abdominal pain using the standard 10-cm visual analogue scale (VAS). VAS score is evaluated between 0 to 10, higher score means worse pain.

SECONDARY OUTCOMES:
Stress hormone response | 5 hours
  Blood is going to be taken and recorded in a yellow capped gel biochemistry tube (SSTM II Advance Tubes) for the measurement of stress hormone glucose (70-100mg/dl), prolactin (4.79-23.3µg/dl), cortisol (60.2-184µg/dl) 1 hour before and 1 hour after the operation
Analgesia period | 24 hours
  The time from the end of the operation to the first analgesic requirement was determined as the "analgesic period" and this time is going to be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No